CLINICAL TRIAL: NCT06966271
Title: Investigation of the Relationship Between the Respiratory Profile of Patients With Obstructive Pulmonary Disease and the Effectiveness of the Inhalation Therapies
Brief Title: Investigation of the Respiratory Profile of Patients With Obstructive Pulmonary Disease (ASTHMA, COPD)
Acronym: OPTIPULM
Status: Recruiting | Type: Observational
Sponsor: Tradeflex Ltd (Industry)
Collaborators: Medisol Development Kft. (Industry)
Responsible Party: Sponsor
Other Study IDs: NNGYK/GYSZ/36422-4/2024
Record Dates: First submitted 2025-05-02; First posted 2025-05-11 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Asthma Bronchiale; COPD
Keywords: inhalation therapy; computer modelling; aerosol drug delivery
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The primary aim of the OPTIPULM study is the evaluation of recorded pulmonary function curves and, based on them, the computer modelling of lung deposition for the individually used or potentially applicable inhalation drugs. The secondary aims include assessing the patients' inhalation device usage and providing recommendations for its optimization based on the recorded breathing curves and deposition calculations. The study also compares results across different flow rates and device resistances, aiming to identify the device with the highest modelled lung deposition for each patient.

Understanding and Improving Inhalation Therapy in Lung Disease The OPTIPULM study looks at how well inhaled medications reach the lungs of people living with asthma or COPD (chronic obstructive pulmonary disease). It aims to improve treatment by helping doctors choose the best inhaler for each patient based on how they breathe.

Every patient breathes differently, and not all inhalers work the same way. Sometimes the medicine doesn't reach deep enough into the lungs, which can make treatment less effective. This study helps doctors better understand which device works best for each individual.

What happens during the study? No new treatments or changes to medication are made.

Patients do a regular breathing test (like blowing into a tube). A computer program uses this breathing data to simulate how much medicine reaches the lungs with different inhalers.

Doctors can then make more personalized choices for inhalation therapy.

Who can take part? Adults with asthma or COPD who are able to use their inhaler correctly and complete a breathing test.

What is the benefit? Although the study does not change treatments directly, it helps improve future care by identifying the best-matching inhaler for each patient. This can lead to better symptom control and fewer exacerbations.

DETAILED DESCRIPTION:
Study Title:

Assessment of the Relationship Between Inhalation Therapy Effectiveness and Breathing Profiles in Patients with Obstructive Pulmonary Diseases (OPTIPULM)

The primary goal of this observational cross-sectional study is to analyze the relationship between patients' breathing characteristics and the effectiveness of their inhaled therapies. The study targets adult patients diagnosed with asthma or chronic obstructive pulmonary disease (COPD).

Background and Rationale:

Asthma and COPD are chronic obstructive airway diseases with increasing prevalence worldwide. Despite the availability of a wide range of inhaled medications and delivery devices, therapy is often suboptimal due to patient-specific factors such as improper inhalation technique or mismatch between inhaler resistance and the patient's inspiratory capacity.

Emerging data suggest that aerosol deposition in the lungs-and therefore the efficacy of treatment-can be significantly influenced by the individual's breathing profile and the inhalation device used. However, this is rarely taken into account in routine clinical practice.

Study Objectives:

Primary Objective:

To evaluate individual pulmonary function test (PFT) data and, based on this, to model and estimate drug deposition in the lungs using computer simulation for various inhaler-drug combinations.

Secondary Objectives:

To assess the inhalation techniques of patients.

To recommend device optimization strategies based on flow-resistance matching.

To identify which device (among commercially available options) is most likely to deliver the highest lung deposition for the individual patient.

ELIGIBILITY:
Primary Outcome Measure:

Estimated Lung Deposition of Inhaled Medication (% of Emitted Dose): The proportion of the inhaled drug dose predicted to deposit in the lungs, calculated via computer modeling using each participant's individual pulmonary function curve and inhalation parameters.

Inclusion criteria:

* Diagnosed obstructive pulmonary disease (asthma or COPD) confirmed by a pulmonologist.
* Proper use of inhalation device after training.
* Routine pulmonary function test performed during medical visit.
* Ambulatory (non-hospitalized) patient.
* Age over 18 years.
* Mentally competent and able to consent.

Exclusion criteria:

* Failure to meet any of the inclusion criteria.
* Inability to complete the relevant parts of the questionnaire.
* Refusal to consent to participation.
* Presence of untreated severe chronic illness.
* Invalid or improperly conducted pulmonary function test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes adult outpatients (≥18 years old) diagnosed with obstructive airway diseases, specifically asthma or chronic obstructive pulmonary disease (COPD). Patients must be under the care of a pulmonologist and capable of performing a routine pulmonary function test (spirometry). Participants are required to demonstrate the correct use of their prescribed inhaler following brief education and instruction.
  The population may include a range of disease severities (mild to severe) and treatment regimens, reflecting real-world inhaler usage. Both male and female participants are eligible, with no restriction on ethnicity or socioeconomic status. Participants must be mentally competent and able to provide informed consent.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Correlation of respiratory function with inhalation drug deposition deposition | 01.01.2025 - 30.07.2025
  The aims of the study are to evaluate the recorded respiratory function (spirometry), and on this basis, computer modelling of the lung deposition of inhalation drugs and selection of personalised therapy.

CONTACTS AND LOCATIONS:
Overall Officials: János Varga, Prof., Principal Investigator — Semmelweis University
Locations (7):
- Hungary (7):
  - Országos Korányi Pulmonológiai Intézet, Budapest
  - Csornai Margit Kórház Pulmonológiai és Allergológia Szakambulancia, Csorna
  - Debreceni Egyetem Tüdőgyógyászati Klinika, Debrecen
  - Dunakeszi-SZTK Nonprofit Kft. Tüdőgyógyászat, Dunakeszi
  - Győr-Moson-Sopron Vármegyei Petz Aladár Egyetemi Oktató Kórház, Győr
  - • Szegedi Tudományegyetem Szent-Györgyi Albert Klinikai Központ Tüdőgyógyászati Klinika, Szeged
  - Református Pulmonológiai Centrum, Törökbálint

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Horvath A, Farkas A, Szipocs A, Tomisa G, Szalai Z, Galffy G. Numerical simulation of the effect of inhalation parameters, gender, age and disease severity on the lung deposition of dry powder aerosol drugs emitted by Turbuhaler(R), Breezhaler(R) and Genuair(R) in COPD patients. Eur J Pharm Sci. 2020 Nov 1;154:105508. doi: 10.1016/j.ejps.2020.105508. Epub 2020 Aug 21. PMID 32836137